CLINICAL TRIAL: NCT06072807
Title: Brain [18F]-FES PET/CT in the Diagnosis, Treatment Planning and Response Assessment of Brain Metastases in Patients With Estrogen-Receptor Positive Breast Cancer
Brief Title: Brain [18F]-FES PET/CT in Patients With Estrogen-Receptor Positive Breast Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-02025733
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Brain Metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ER Positive Breast Cancer Patients with Brain Metastases (Experimental): A diagnostic intervention where this group will undergo an additional 18F- FES PET/CT scan in addition to their standard of care MRI and FDG PET/CT scan.
  Interventions: Diagnostic Test: Brain Imaging with 18F-FES

INTERVENTIONS:
Diagnostic Test: Brain Imaging with 18F-FES — Using 18F-FES radiotracer in PET/CT scan to evaluate brain metastases in ER positive breast cancer patients.

SUMMARY:
The goal of this interventional study is to optimize the protocol of FES PET/CT in Estrogen Receptor positive Breast cancer patients with Brain metastases. Patients will undergo MRI of the brain and FDG PET/CT brain as part of standard of care for radiation treatment planning. An additional 18F-FES PET/CT brain scan will be completed before this standard of care radiation treatment. Patients will be followed prospectively with clinical and MRI assessments per standard-of-care for a total of 12 months.

Study Population: Patients with ER-positive breast cancer with biopsy proven or suspected new or recurrent brain metastases (based on standard of care MRI) planned for radiation treatment of brain lesions.

DETAILED DESCRIPTION:
Objectives

1. Evaluate the kinetics of dynamic brain FES PET/CT and optimize acquisition protocol.
2. Evaluate utility of FES PET/CT as an adjunct modality in radiotherapy planning.
3. (Exploratory aim) Determine correlation between FES PET metrics and survival metrics.

Overall Design All subjects will undergo a MRI brain and FDG PET/CT brain scan as part of clinical standard- of-care for radiation treatment planning. An additional 18F-FES PET/CT brain scan will be performed as part of this study prior to standard of care radiation treatment. 18F-FES is clinically approved for the study population, however has to date not been widely used in the clinical context of differentiating brain metastases from radiation sequela. The 18F-FES PET/CT scan will be completed within approximately 2 days to 4 weeks of the 18F-FDG PET/CT, and 2 days to 4 weeks of the MRI brain, respectively. While MRI and PET can be performed on the same day if needed, the 18F-FDG PET/CT and 18F-FES PET/CT have to be separated by at least 1 day, to allow for 10 half-lives of 18F (10 times 108 minutes = 18 hours) to pass in order to avoid signal overlap on the second PET/CT scan. Subjects will be followed prospectively with clinical and MRI assessments per clinical standard-of-care for a total of 12 months.

Aim 1

* 5 mCi FES +/- 10% will be injected intravenously (per manufacturer's recommendations). FES PET/CT will be obtained in dynamic 3D list mode for 90 minutes starting from injection.
* Kinetic analysis of dynamic PET images will be carried out using a reversible 1-tissue-2- compartment model as well as Logan Vt, and the influx rate constant, Ki, and distribution volume, Vt, will measured respectively.
* Static 10min PET images will be generated for from 50 to 80 min on a 10min increment, and the corresponding SUV's and tumor-to-background ratios will be compared to that in the 80- 90min imageset, a workflow that previously established by our group using DOTATATE PET/MR in meningioma, and using FLT/FMISO PET/CT in high-grade glioma.
* Tumor volume will be delineated using PMOD (PMOD, Zurich), a dedicated tool for PET analyses and kinetic modeling.

Aim 2.

* To evaluate utility of FES PET/CT in RT planning, planning treatment volumes will be delineated by a radiation oncologist in conjunction with a neurosurgeon based on MRI (gold standard); subsequently, the FES PET/CT data will be made available to the radiation oncologist, and the planning treatment volume (PTV) will be modified accordingly if necessary.
* The clinical treatment plan will be modified (as a proof-of-concept) based on the MRI+FES PTV, and the target dose volume histograms (DVH) will be compared to the MRI-based (gold standard).
* Change in management based on additional information provided in the PET data will be recorded. In an exploratory analysis, FES PET will be compared with standard of care FDG PET/CT or PET/MR for treatment planning.

ELIGIBILITY:
Inclusion Criteria:

1. Active diagnosis of ER+ breast cancer (biopsy proven) and new or recurrent brain metastases (biopsy proven or suspected based on MRI appearance)
2. Ability to provide informed consent
3. Discontinuation of ER modulators for at least 8 weeks, and discontinuation of ER down regulators for at least 28 weeks (as per manufacturer guidelines)
4. Age >=18 years
5. Eastern Cooperative Oncology Group performance score 0-1
6. Life expectancy >=6 months
7. Planned for radiation treatment for brain metastases

Exclusion Criteria:

1. Pregnancy
2. Unable to undergo Standard of Care
3. Allergy to FES.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean SUV | 3 years
  Mean standardized uptake value within a region of interest placed based on MRI findings of suspicious brain lesion.
Maximum SUV | 3 years
  Maximum standardized uptake value within a region of interest placed based on MRI findings of suspicious brain lesion.
SUV Ratio | 3 years
  Standardized uptake value ratio of target lesion over reference region.
Target-to-Background Ratio | 3 years
  Qualitative appearance of lesion delineation on PET.
Influx (Ki) | 3 years
  Parametric PET analysis results within the same region of interest as that for Maximum SUV.
Distribution volume (Vt) for scan times | 3 years
  Distribution volume (Vt), measured within the same region of interest as that for Maximum SUV, for scan times ranging between 45 min and 85 min with 5min intervals and corresponding results will be compared to those measured with the full dataset at 90mm.

SECONDARY OUTCOMES:
Proportion of cases in which there was a change in management based on FES PET/CT | 3 years
  We will compare RT plans devised based on contrast-enhanced brain MRI alone (gold standard) to RT plans incorporating FES PET/CT as an adjunct modality and will quantify the proportion of cases in which there was a change in management based on FES PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Ivanidze, MD/PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York-Presbyterian/Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No